CLINICAL TRIAL: NCT00762047
Title: Phase 2 IDE Study of Durasphere FI in the Treatment of Fecal Incontinence
Brief Title: A Prospective, Multi-center, Randomized, Blinded Study to Evaluate Durasphere FI for the Treatment of Fecal Incontinence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Carbon Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P1004
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2012-01

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Durasphere (Experimental)
  Interventions: Device: Durasphere FI
- Sham (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: Durasphere FI — Durasphere Injection
  Arms: Durasphere
Device: Sham — Sham injection with anesthesia
  Arms: Sham

SUMMARY:
The purpose of this study is to evaluate a new injectable bulking agent for the treatment of fecal incontinence in adult men and women. This study has been designed to assess the safety, effectiveness and performance of Durasphere in adults suffering from fecal incontinence under monitored clinical conditions.

The frequency and severity of fecal incontinence symptoms will be measured using a modified Cleveland Clinic Incontinence Score as the primary criteria by which success is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* History of fecal incontinence;
* Incontinence episodes over a 14-day period;
* Eighteen years of age or older;

Exclusion Criteria:

* Abnormalities of the external sphincter greater than 10 mm;
* Fibrosis of the tissue at the likely injection sites;
* Has a condition that could lead to significant postoperative complications
* Rectal varices;
* Cancer of the rectum or colon, undergoing active treatment;
* Crohn's disease or ulcerative colitis;
* Chronic diarrhea unmanageable by drugs and/or diet;
* Rectal bleeding;
* Pregnant or within one year postpartum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-06; Primary Completion 2008-08 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The frequency and severity of fecal incontinence symptoms will be measured using a modified Cleveland Clinic Incontinence Score | 6 month
Safety will be demonstrated through an analysis of morbidity and complication rates associated with Durasphere. | Throughout study
The proportion of patients maintaining a 25% improvement in Cleveland Clinic Incontinence Score | 12 month

REFERENCES:
- See also: Related Info — http://carbonmed.com